CLINICAL TRIAL: NCT06785298
Title: Clinical Study to Evaluate the Possible Efficacy and Safety of Fexofenadine in Patients With Parkinson's Disease Treated With Conventional Treatment
Brief Title: Fexofenadine as Adjuvant Therapy in Parkinson Disease
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ihab Elsayed Hassan, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3245
Record Dates: First submitted 2024-11-25; First posted 2025-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Fexofenadine
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; fexofenadine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control arm (Active Comparator): will receive their standard dopamine replacement therapy for 6 months.
  Interventions: Drug: Levodopa/carbidopa
- Fexofenadine group (Active Comparator): will receive Fexofenadine 180 mg once daily together with their standard dopamine replacement therapy for 6 months
  Interventions: Drug: Levodopa/carbidopa; Drug: Fexofenadine

INTERVENTIONS:
Drug: Levodopa/carbidopa — A dopamine precursor, was first developed for the treatment of PD in the 1960s and continues to be the most-effective therapeutic agent for PD
Drug: Fexofenadine — Fexofenadine is a second-generation antihistamine that does not penetrate the CNS and has the least CNS side effects among the second-generation antihistamines
  Arms: Fexofenadine group

SUMMARY:
Parkinson's disease (PD) is a chronic, progressive neurological disorder characterized by both motor and non-motor symptoms. PD is the second most common neurodegenerative disorder after Alzheimer's disease and the most common movement disorder. PD has age-related pathology; it is present in 1-2% of the population over 60 years of age. The disease is characterized by a triad of disordered voluntary motor activity in the form of bradykinesia (slowness of movement) or even akinesia (absence of movement),rigidity and postural instability, and a resting tremor of the hands and less commonly the feet.

ELIGIBILITY:
Inclusion Criteria:• Age ≥ 50 years. Both male and female will be included. Patients with Parkinson's disease on dopamine replacement therapy. Modified Hoehn and Yahr stage, MHY 1-4

Exclusion Criteria:• Atypical parkinsonism or drug-induced parkinsonism Breast feeding Pregnant women and women with planned pregnancy. Patients with significant liver and kidney function abnormalities. History/presence of acute heart disease Alcohol and / or drug abusers. Patients with known allergy to the study medications Other medical conditions that can interfere with results or endanger the participant.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the change in quality of life in Parkinson's disease by Unified Parkinson's Disease Rating Scale | 6 months
  The primary outcome is the change in quality of life in Parkinson's disease by Unified Parkinson's Disease Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt